CLINICAL TRIAL: NCT03869632
Title: First in Human Dose Escalation Study of YL-13027 Monotherapy in Subjects With Advanced Stage Solid Tumors
Brief Title: First in Human Dose Escalation Study of YL-13027 in Subjects With Advanced Stage Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai YingLi Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YL-13027-001
Record Dates: First submitted 2019-03-08; First posted 2019-03-11 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Advanced Solid Tumors
Keywords: YL-13027; Advanced Solid Tumors

STUDY DESIGN:
Intervention Model Description: dose escalation
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- YL-13027 (Experimental): YL-13027 tablets will be given daily for 28 days in 28-day cycles until there appears evidence of progressive disease, intolerable toxicity, or the subject discontinues from the study treatment for other reasons.
  Interventions: Drug: YL-13027

INTERVENTIONS:
Drug: YL-13027 — Daily doses by oral administration on each day of each 28 day cycle. Starting dose is 60mg, with escalation to 360mg, and subsequent dose escalation using a modified Fibonacci algorithm.

SUMMARY:
YL-13027-001 is a phase I open-label, first in human, dose escalation study which investigate the tolerability, safety, pharmacokinetics (PK) and efficacy of YL-13027 in subjects with advanced stage solid tumors.

DETAILED DESCRIPTION:
This is a open-label, single-center, dose-escalation, phase I study of YL-13027 comprised of a dose escalation part and a dose expansion part in subjects with advanced stage solid tumors. The study will investigate the tolerability, safety, pharmacokinetics (PK) and efficacy of YL-13027, and will define the maximum tolerated dose (MTD) of YL-13027 using an accelerated titration test and 3+3 design. a dose expansion part will identify the recommended phase 2 dose. YL-13027 is an orally bioavailable small molecule that inhibits protein serine/threonine kinase of activin receptor-like kinase 5 (ALK5) and blocks intracellular signaling of TGF-β by inhibiting the phosphorylation of ALK5 substrates. In this clinical trial, YL-13027 is given orally daily. A treatment cycle is defined as 28 days. Adverse events (AEs) were graded by NCI-CTCAE V5.0. Efficacy was evaluated according to RECIST V1.1.

ELIGIBILITY:
Inclusion Criteria:

1. Males and/or females age from 18 to 75;
2. Histologically or cytologically confirmed patients with advanced malignant solid tumors, eligible patients must have failed standard treatment, no standard treatment, or not suitable for standard treatment at this stage as determined by the investigator;
3. In the dose escalation portion, both measurable and non-measurable tumor lesions were acceptable according to RECIST1.1 criteria;There was at least one measurable tumor lesion in the dose expansion portion;
4. Eastern Cooperative Oncology Group performance status of 0 to 1;
5. Life expectancy of at least 3 months;
6. Acceptable organ function: Absolute neutrophil count(ANC)≥1.5×109/L; Platelet count(PLT)≥100×109/L; Hemoglobin(Hb)≥90 g/L; Total bilirubin(TBIL)≤1.5×Upper limit of normal value(ULN); Alanine aminotransferase(ALT)≤2.5×ULN; Aspartate aminotransferase(AST)≤2.5×ULN; Creatinine(Cr)≤1.5×ULN; Creatinine clearance ≥50ml/min;Left Ventricular Ejection Fractions(LVEF)≥50%； QTcF<450 ms;
7. The washout period from the last time accepting any anti-tumor treatment (including radiation therapy, chemotherapy, hormone therapy, surgery, or molecular targeted therapy) to participating in this test should be 3 weeks or more.The washout period of oral fluorouracil should be 2 weeks or more, and that of mitomycin and nitrosocarbamide should be 6 weeks or more;
8. Fertile male and female must agree to use medically approved contraceptives during the study and within 6 months after the last dose of the study;
9. Female who is capable of conceiving:Blood pregnancy tests should be negative 7 days before the first dose; Patients cannot breastfeed, if the subject has stopped breastfeeding at the time of study entry, the cessation of breastfeeding must be from the day of first dose to more than 30 days after the last dose;
10. The last time participate in an investigational drug study should be more than one month prior to the study entry;
11. According to the judgment of the investigator, the subject has high compliance and is willing to complete the experiment and comply with the protocol;
12. Voluntary participation in this clinical trial, understanding of the study procedures and the ability to sign informed consent forms (ICFs).

Exclusion Criteria:

1. There are third interstitial effusions (such as massive pleural effusion and ascites) which can not be controlled by drainage or other methods;
2. Within 3 months before the first dose, grade 3 or grade 4 gastrointestinal bleeding or varicose bleeding and requiring blood transfusion or endoscopic or surgical intervention has happened;
3. Medical history of difficulty in swallowing, malabsorption, or other chronic gastrointestinal disease, or conditions that may hamper compliance and/or absorption of the tested product;
4. subjects with a definitely history of neurological or psychiatric disorders;
5. Known infection with human immunodeficiency virus (HIV), hepatitis B virus(HBV), or hepatitis C virus (HCV);
6. History of immunodeficiency, including HIV positive test, other acquired or congenital immunodeficiency disorders, organ transplantation or allogeneic bone marrow transplantation;
7. Exists moderate or severe heart disease: (1) Within 6 months before the first dose,myocardial infarction, angina, grade III/IV congestive heart failure, pericardial effusion, uncontrollable severe hypertension (up to 150/90 mmHg or less) (2) ECG abnormalities with clinical significance: symptomatic or persistent atrial or ventricular arrhythmias, degree II or III atrioventricular block, bundle branch block, ventricular hypertrophy; (3) The echocardiogram shows significant abnormalities: For example, moderate or severe heart valve function defects are assessed according to the normal lower limit of the institution;Patients with minor or mild valve regurgitation (tricuspid, pulmonary, mitral, or aortic) can be included in this study (4) Laboratory examination shows brain natriuretic peptide or troponin T levels increases (5) Various factors that may increase the risk of QTcF prolonging or arrhythmia events. For example, hypokalemia, congenital long QT syndrome, may prolong the QT interval of various combined drugs, etc. (6) Predisposition factors cause the development of ascending aorta or aortic arch aneurysm: For example, marfan syndrome, CT records of the history of cardiac vascular injury; (7) History of heart or aortic surgery.
8. Patients with central nervous system metastasis;
9. At the beginning of the study, the unrecovered toxicity of the previous treatment exceeded CTCAE5.0 grade 1(except for hair loss);
10. Previously treated with TGF-β inhibitors;
11. According to the judgement of the researcher,there are concomitant diseases that seriously endanger the safety of patients or affect the completion of the study (such as severe hypertension, diabetes, thyroid diseases, etc.).
12. subjects, in the opinion of the the Investigator, who are unsuitable to participate in the study for any other reason.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2019-03-19 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Dose limited toxicities evaluated with NCI-CTC AE v5.0 | within 28 days after the first dose
  Incidence of dose limited toxicities and associated dose of YL-13027
Adverse events evaluated by NCI CTCAE v5.0 | from the first dose to within 30 days after the last dose
  Incidence of adverse events and associated dose of YL-13027

SECONDARY OUTCOMES:
Plasma concentration of YL-13027 | within 56 days after the first dose
  This composite endpoint will measure the plasma concentration of YL-13027
Objective response rate | within 30 days after the last dose
  the proportion of subjects who have a Complete Response or Partial Response
Disease control rate | within 30 days after the last dose
  the proportion of subjects who have a Complete Response or Partial Response

CONTACTS AND LOCATIONS:
Overall Officials: Hanying Bao, PhD, Study Director — Shanghai YingLi Pharmaceutical Co. Ltd.
Locations (1):
- Shanghai East Hospital, Shanghai, Shanghai Municipality, China